CLINICAL TRIAL: NCT00436306
Title: Stage Matched Intervention to Increase Dual Method Use
Acronym: PROTECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Peipert, Robert J. Terry Professor, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD036663 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Contraception; Sexually Transmitted Diseases; Pregnancy
Keywords: prevention; behavior; risk reduction behavior
MeSH Terms: conditions — Sexually Transmitted Diseases; Behavior; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized Intervention: stage-matched/tailored counseling (Experimental): Individualized Intervention is a computer-based, stage-matched, tailored intervention to promote the use of dual methods of contraception for STD and unplanned pregnancy prevention.
  Interventions: Behavioral: Individualized Intervention; Behavioral: Computer-based contraceptive information
- Control: Enhanced usual care counseling (Placebo Comparator): The Enhanced Usual Care arm was the control group. It provided computer-based information regarding contraceptive methods, but was not individualized or tailored to the participant stage of change.
  Interventions: Behavioral: Computer-based contraceptive information

INTERVENTIONS:
Behavioral: Individualized Intervention — Individualized Intervention is a computer-based, stage-matched, tailored intervention to promote the use of dual methods of contraception for STD and unplanned pregnancy prevention.
  Arms: Individualized Intervention: stage-matched/tailored counseling
Behavioral: Computer-based contraceptive information — Contraceptive method information is provided on a computer.

SUMMARY:
The primary purpose of Project PROTECT was to evaluate two different intervention approaches that encourage young women to use dual methods of contraception. The individualized intervention is a computer assisted, fully-tailored, interactive intervention based on the transtheoretical model of behavior change. This intervention was compared to an enhanced standard care intervention that provided computer-based, non-tailored information and advice regarding the use of contraceptive methods. The two primary outcomes of this trial include: 1) a behavioral outcome: the reported use of dual methods of contraception; and 2) a biological outcome: an incident or recurrent STI or unintended pregnancy. The hypotheses of this trial were: 1) the individualized intervention will result in a greater increase in dual contraceptive use than the standard care approach; and 2) the individualized intervention would result in greater protection against incident or recurrent cases of sexually transmitted infections and unplanned pregnancies.

DETAILED DESCRIPTION:
Protection from both sexually transmitted infections (STIs), human immunodeficiency virus (HIV), and unintended pregnancy can be achieved with the use of dual methods of contraception. This proposal was designed to develop, implement, and evaluate the impact of an innovative, computer-assisted stage-based individualized interactive intervention (Individualized Intervention) based on the transtheoretical compared to enhanced standard care counseling on the use of dual methods of contraception. Primary outcomes, including behavioral and biological outcomes, were assessed in this randomized clinical trial of 550 high-risk women. Participants were followed at 6 month intervals for 24 months with follow-up interviews to determine reported use of dual methods of contraception (behavioral outcome). Clinical examinations at 12 and 24 months and with new onset of symptoms assessed biological outcomes including incident or recurrent cases of STI and unintended pregnancy. Secondary outcomes included intermediate outcome variables such as changes in stage of change, processes of change, decisional balance, and self-efficacy. The primary hypotheses of this study were: 1. the Individualized Intervention will result in increased dual contraceptive use; 2. the Individualized Intervention will result in protection against new cases of STIs, re-infection with sexually transmitted organisms, and unplanned pregnancies; and 3. the Individualized Intervention will lead to the greatest changes in secondary outcome measures. If found to be effective, the stage-matched intervention has potential for widespread dissemination in schools, clinics, offices, and community centers to prevent STIs/HIV and unintended pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. Sexually active with a male partner in the past 6 months
3. Desire to avoid conception for 24 months or more
4. High risk for unintended pregnancy or STI:

   * Age less than 25
   * Age 25 and older with:

     * History of unplanned pregnancy
     * History of a sexually transmitted infection
     * Inconsistent use of contraception
     * Other factors felt to place a patient at above average risk for unplanned pregnancy or STI

Exclusion Criteria:

1. currently using dual methods of contraception consistently and correctly.
2. incompetent or unable to give consent;
3. currently pregnant or desires pregnancy in the next 24 months.

Ages: 13 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 550 (Actual)
Dates: Start 1999-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Behavioral: reported use of dual methods of contraception | 24 months
  Outcome: ANY use of dual methods of contraception.
  Also evaluated consistent condom use.
Biological: incident sexually transmitted infection or unintended pregnancy | 24 months
  ANY sexually transmitted infection OR unintended pregnancy.

SECONDARY OUTCOMES:
Secondary outcomes will include intermediate outcomes variables such as | 24 months
  Secondary outcomes: ANY sexually transmitted infection; unplanned pregnancy; incident infection with Chlamydia trachomatis, Neisseria gonorrhoeae, Trichomonas vaginalis, or pelvic inflammatory disease.
changes in stage of change, processes of change, decisional balance, and self-efficacy. | 24 months
  Advancement through the stages of change, and changes in the processes of change, decisional balance, and self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Peipert, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Peipert J, Redding CA, Blume J, Allsworth JE, Iannuccillo K, Lozowski F, Mayer K, Morokoff PJ, Rossi JS. Design of a stage-matched intervention trial to increase dual method contraceptive use (Project PROTECT). Contemp Clin Trials. 2007 Sep;28(5):626-37. doi: 10.1016/j.cct.2007.01.012. Epub 2007 Feb 7. PMID 17374567
- [Result] Matteson KA, Peipert JF, Allsworth J, Phipps MG, Redding CA. Unplanned pregnancy: does past experience influence the use of a contraceptive method? Obstet Gynecol. 2006 Jan;107(1):121-7. doi: 10.1097/01.AOG.0000192170.16746.ea. PMID 16394049
- [Result] Peipert JF, Lapane KL, Allsworth JE, Redding CA, Blume JL, Lozowski F, Stein MD. Women at risk for sexually transmitted diseases: correlates of intercourse without barrier contraception. Am J Obstet Gynecol. 2007 Nov;197(5):474.e1-8. doi: 10.1016/j.ajog.2007.03.032. Epub 2007 Aug 21. PMID 17714677
- [Result] Peipert JF, Lapane KL, Allsworth JE, Redding CA, Blume JD, Stein MD. Bacterial vaginosis, race, and sexually transmitted infections: does race modify the association? Sex Transm Dis. 2008 Apr;35(4):363-7. doi: 10.1097/OLQ.0b013e31815e4179. PMID 18360319
- [Result] Krings KM, Matteson KA, Allsworth JE, Mathias E, Peipert JF. Contraceptive choice: how do oral contraceptive users differ from condom users and women who use no contraception? Am J Obstet Gynecol. 2008 May;198(5):e46-7. doi: 10.1016/j.ajog.2007.12.025. Epub 2008 Mar 7. PMID 18313637
- [Result] Peipert JF, Redding CA, Blume JD, Allsworth JE, Matteson KA, Lozowski F, Mayer KH, Morokoff PJ, Rossi JS. Tailored intervention to increase dual-contraceptive method use: a randomized trial to reduce unintended pregnancies and sexually transmitted infections. Am J Obstet Gynecol. 2008 Jun;198(6):630.e1-8. doi: 10.1016/j.ajog.2008.01.038. Epub 2008 Apr 8. PMID 18395692
- [Result] Kuroki LM, Allsworth JE, Redding CA, Blume JD, Peipert JF. Is a previous unplanned pregnancy a risk factor for a subsequent unplanned pregnancy? Am J Obstet Gynecol. 2008 Nov;199(5):517.e1-7. doi: 10.1016/j.ajog.2008.03.049. Epub 2008 May 12. PMID 18468575
- [Result] Allsworth JE, Anand M, Redding CA, Peipert JF. Physical and sexual violence and incident sexually transmitted infections. J Womens Health (Larchmt). 2009 Apr;18(4):529-34. doi: 10.1089/jwh.2007.0757. PMID 19245303
- [Result] Allsworth JE, Peipert JF. Severity of bacterial vaginosis and the risk of sexually transmitted infection. Am J Obstet Gynecol. 2011 Aug;205(2):113.e1-6. doi: 10.1016/j.ajog.2011.02.060. Epub 2011 Feb 27. PMID 21514555
- [Result] Peipert JF, Zhao Q, Meints L, Peipert BJ, Redding CA, Allsworth JE. Adherence to dual-method contraceptive use. Contraception. 2011 Sep;84(3):252-8. doi: 10.1016/j.contraception.2011.01.023. Epub 2011 Apr 16. PMID 21843690